CLINICAL TRIAL: NCT06280495
Title: Neoadjuvant Combination of Serplulimab and Bevacizumab With FOLFOX Versus FOLFOX Alone for Resectable Liver Metastases in RAS/BRAF Wild-Type, pMMR/MSS Colorectal Cancer Patients
Brief Title: Neoadjuvant Serplulimab & Bevacizumab With FOLFOX vs. FOLFOX Alone in RAS/BRAF WT, pMMR/MSS CRC Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTENSIFY-CRC
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; spartalizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, multicenter clinical trial. Stratified randomization based on liver metastasis characteristics, including timing, number, and size, will be conducted in eligible patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFOX only group (Active Comparator): Oxaliplatin: 85 mg/m2 IV on day 1 Fluorouracil (FU): 400 mg/m2 IV bolus on day 1, followed by 2.4 g/m2 continuous IV infusion over 48 hours Leucovorin: 200 mg/m2 IV on day 1 This treatment regimen is repeated every two weeks for a total of 6 cycles.
  Interventions: Drug: Oxaliplatin; Drug: Fluorouracil
- Serplulimab + Bevacizumab + FOLFOX (Experimental): Serplulimab: 200 mg IV infusion on day 1 Bevacizumab: 5 mg/kg IV infusion on day 1 Oxaliplatin, FU, and Leucovorin as per the control arm The experimental arm follows the same treatment schedule as the standard FOLFOX regimen, with the addition of Serplulimab and Bevacizumab for the first 3 cycles only.
  Interventions: Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Serplulimab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Oxaliplatin — 5 mg/m2 IV on day 1
  Other Names: Eloxatin
Drug: Fluorouracil — 400 mg/m2 IV bolus on day 1, followed by 2.4 g/m2 continuous IV infusion over 48 hours
  Other Names: 5-FU
Drug: Serplulimab — 200 mg IV infusion on day 1
  Other Names: anti-PD-1 antibody
  Arms: Serplulimab + Bevacizumab + FOLFOX
Drug: Bevacizumab — 5 mg/kg IV infusion on day 1
  Other Names: Avastin
  Arms: Serplulimab + Bevacizumab + FOLFOX

SUMMARY:
The primary objective of this study is to assess whether the addition of Serplulimab (a PD-1 inhibitor) and Bevacizumab (an anti-angiogenesis agent) to the standard FOLFOX chemotherapy can enhance the immune microenvironment in the liver, increase T lymphocyte infiltration, and consequently improve the postoperative prognosis for patients with surgically resectable colorectal cancer liver metastases (RAS/BRAF wild-type, pMMR/MSS) compared to FOLFOX alone.

DETAILED DESCRIPTION:
In this prospective, multi-center clinical trial titled "INTENSIFY," we seek to evaluate the potential benefits of integrating Serplulimab and Bevacizumab with the standard FOLFOX chemotherapy regimen as neoadjuvant treatment for surgically resectable colorectal cancer liver metastases (CRLM). Colorectal cancer remains a leading cause of global cancer-related morbidity and mortality, with liver metastases accounting for a significant proportion. Our primary objective is to investigate whether the addition of Serplulimab, a PD-1 inhibitor, and Bevacizumab, an anti-angiogenesis agent, can improve the postoperative prognosis for patients with RAS/BRAF wild-type, pMMR/MSS CRLM. We aim to address critical questions regarding the efficacy of this combined treatment in enhancing the immune microenvironment within the liver, ultimately leading to increased T lymphocyte infiltration and improved patient outcomes. The study will involve a randomized assignment of patients to either the standard FOLFOX chemotherapy arm or the experimental arm receiving FOLFOX in combination with Serplulimab and Bevacizumab. Participants will undergo neoadjuvant treatment, surgical resection, and regular follow-up assessments to evaluate treatment response, recurrence rates, and overall survival. By comparing outcomes between the two groups, specifically assessing factors like recurrence-free survival, overall survival, and changes in the immune microenvironment, we aim to provide valuable insights into the optimization of treatment strategies for this specific subset of colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old
* Histologically confirmed colorectal adenocarcinoma
* Radiological and/or pathological confirmation of liver metastases, with ≤5 lesions
* Genetic testing and/or immunohistochemistry confirmation of RAS, BRAF wild-type, and pMMR/MSS
* Absence of extrahepatic metastases confirmed by CT, MRI, or PET/CT (if necessary)
* Primary colorectal tumor has been or can be radically resected
* Liver metastatic lesions are resectable (including radiofrequency ablation and SBRT), and postoperative NED (no evidence of disease) is expected. Resectable liver metastases are specifically defined as ① ≤5 metastatic lesions; ② R0 resection can be performed (including radiofrequency ablation and SBRT); ③ Sufficient residual liver volume is expected after resection; ④ At least one hepatic vein can be preserved after resection, with preserved blood flow in and out of the residual liver and preserved bile ducts, and can preserve at least two adjacent liver segments; ⑤ No extrahepatic metastases.
* No prior anti-tumor therapy for liver metastases, except for surgical resection of primary lesions
* Normal hematological function (platelets >90×109/L; white blood cells >3×109/L; neutrophils >1.5×109/L)
* Serum bilirubin ≤1.5 times the upper limit of normal (ULN), transaminases ≤5 times ULN, alkaline phosphatase ≤2.5 ULN, no ascites, normal coagulation function, albumin ≥35g/L
* Liver function classified as Child-Pugh grade A
* Serum creatinine below the upper limit of normal (ULN), or calculated creatinine clearance rate >50ml/min (using Cockcroft-Gault formula)
* ECOG performance status 0-1
* Expected lifespan >3 months
* Signed written informed consent
* Willing and able to be followed up until death or end of study or study termination.

Exclusion Criteria:

* Diagnosis of colorectal cancer with distant extrahepatic metastases
* Prior chemotherapy, targeted therapy, intervention, or immunotherapy for liver metastases
* No planned surgical resection for liver metastatic lesions
* Received oxaliplatin-containing adjuvant chemotherapy regimen within the past one year
* Any toxicity residuals from previous chemotherapy, excluding alopecia, such as peripheral neuropathy ≥NCI CTC v3.0 grade 2
* Use of immunosuppressive drugs one week prior to study treatment initiation, excluding topical corticosteroids via nasal, inhalational, or other routes or physiological doses of systemic corticosteroids (i.e., not exceeding 10 mg/day of prednisone or equivalent) or steroids used for prevention of contrast agent allergy
* Interstitial lung disease requiring corticosteroid treatment
* Known active autoimmune disease requiring symptomatic treatment or with a history of such disease within the past 2 years. Patients with vitiligo, psoriasis, alopecia, or Graves' disease who have not required systemic treatment within the past 2 years, patients with hypothyroidism requiring only thyroid hormone replacement therapy, and patients with type I diabetes requiring only insulin replacement therapy can be included
* Known history of primary immunodeficiency
* Patients with active tuberculosis
* History of allogeneic organ or hematopoietic stem cell transplantation
* Known allergy to any monoclonal antibody or chemotherapy drug (Fluorouracil, oxaliplatin) preparation or excipient component
* Bleeding tendency or coagulation disorder
* Significant symptoms of intestinal obstruction
* Hypertensive crisis or hypertensive encephalopathy
* Severe uncontrolled systemic complications such as infection or diabetes
* Clinically severe cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), hypertension that remains uncontrolled after appropriate drug treatment, unstable angina pectoris, congestive heart failure (NYHA 2-4), or arrhythmia requiring medication
* Past or physical examination showing central nervous system diseases (such as primary brain tumor, epilepsy uncontrolled by standard treatment, any history of brain metastasis, or stroke)
* Diagnosis of other malignant tumors within the past 5 years (excluding basal cell carcinoma and/or carcinoma in situ of the cervix after radical surgery)
* Patients who received any investigational drug therapy within the last 28 days prior to the study
* Pregnant or lactating women and women of childbearing age not using or refusing to use effective non-hormonal contraception (intrauterine devices, barrier contraception combined with spermicidal gel, or sterilization surgery) or men with reproductive potential unwilling or unable to comply with the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year Progression-Free Survival Rate | Assessed for three years following the initiation of treatment
  The proportion of patients who, following the initiation of treatment, remain both alive and without evidence of disease progression for a consecutive period of three years.

SECONDARY OUTCOMES:
Median Overall Survival | Assessed throughout the study duration (5 years)
  The duration of time from diagnosis until death
Major Pathological Response (MPR) | Assessed following neoadjuvant treatment and resection of CRLM (up to 5 years)
  Defined as residual viable tumor of less than or equal to 10%
Pathologic complete response (pCR) | Assessed following neoadjuvant treatment and resection of CRLM (up to 5 years)
  The absence of tumor cells in all specimens.
Pathological Partial Response | Assessed following neoadjuvant treatment and resection of CRLM (up to 5 years)
  Defined as residual viable tumor of more than 10% but less than 50%
Disease Free Survival | Assessed throughout the study duration (5 years)
  The measure of time after treatment during which no sign of cancer is found
Treatment-related adverse events | Assessed throughout the study duration (5 years)
  Assessment of adverse events related to the treatment received in both arms

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.